CLINICAL TRIAL: NCT06410001
Title: CE-STAND: Cervical Epidural STimulation After Neurologic Damage
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEUROSURG-2023-31800
Record Dates: First submitted 2024-04-19; First posted 2024-05-10 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Spinal Cord Injury
Keywords: Cervical; Spinal cord injury; Epidural spinal cord stimulation; Autonomic dysfunction
MeSH Terms: conditions — Spinal Cord Injuries; Primary Dysautonomias

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Spinal injury patients (Experimental): Experimental: Individuals with cervical SCI comparing stimulation "on" vs "off" longitudinally.
  Interventions: Device: Epidural Spinal Cord Stimulation System

INTERVENTIONS:
Device: Epidural Spinal Cord Stimulation System — Abbott Eterna system implantable pulse generator (IPG), charger, and TriCentrus lead

SUMMARY:
CE-STAND aims to address three areas under-represented in research: chronic, cervical, and autonomic dysfunction. It is both significant and highly impactful, as treating autonomic dysfunction could substantially improve function and quality of life (QoL) in chronic cervical SCI patients.

DETAILED DESCRIPTION:
Spinal cord injury (SCI) affects over 18,000 individuals annually, leading to significant motor and autonomic dysfunctions that reduce quality of life (QoL). Epidural spinal cord stimulation (eSCS) has shown potential in restoring function in chronic individuals with SCI. However, research on cervical, and autonomic dysfunction-related SCI remains limited. This study will assess the safety and efficacy of eSCS in improving autonomic and volitional functions, as well as truncal stability, bowel, bladder, and sexual function, and overall QoL.

The study is a Phase I/II trial in which participants will serve as their own controls. The Abbott Eterna epidural stimulator system will be implanted, and assessments will occur every three months. The study will be conducted over a period of four years. A total of 36 participants will be enrolled and followed for one year.

Bayesian Optimization will be used to determine the most effective stimulation settings, with 15 settings programmed at the end of each visit.

FDA and UMN IRB approvals have been secured for the study. Interim reports will be made available through peer-reviewed journals, conference presentations, and clinical network reporting.

CE-STAND seeks to advance SCI treatment by expanding eSCS applications in chronic cervical SCI, improving patient outcomes, and reducing healthcare costs.

ELIGIBILITY:
Inclusion Criteria:

* Twenty two years of age or older
* Able to undergo the informed consent/assent process
* Stable, motor-complete SCI
* Discrete SCI between C4 and C7 (upper extremity weakness)
* ASIA A or B SCI Classification
* Medically stable in the judgment of the PI
* Intact segmental reflexes below the lesion of injury
* Greater than 1 year since initial injury and at least 6 months from any required spinal instrumentation
* Normal or corrected-to-normal vision to accurately perceive visual stimuli on the N-back task screen, and sufficient hearing ability to accurately perceive auditory stimuli during the task
* Willing to attend all scheduled appointments

Exclusion Criteria:

* Diseases and conditions that would increase the morbidity and mortality of this surgery such as cardiopulmonary.
* Individuals who require respiratory support, including ongoing or intermittent use of a ventilator and/or diaphragmatic pacer
* Inability to withhold antiplatelet/anticoagulation agents perioperatively
* Individuals who have history of recurrent autonomic dysreflexia in the judgment of the PI
* Significant dysautonomia that would prohibit rehabilitation or any history of cerebrovascular accident or myocardial infarction associated with autonomic dysreflexia. A single tilt table test with syncope, presyncope, or SBP < 50 or > 200
* Failure to exhibit cardiovascular autonomic dysfunction on tilt table testing
* Other conditions that would make the subject unable to participate in testing/rehabilitation in the judgment of the PI
* Patients who have participated in another study within the last 12 months in which they have received fluoroscopic or other related radiation exposure
* Current and anticipated need for opioid pain medications or pain that would prevent full participation in the program in the judgment of the PI
* Clinically significant mental illness in the judgment of the PI
* Treatment with botulinum toxin, intrathecal baclofen pump, and antispasmodics will not be permitted unless discussed with and approved by the study PI
* Patients with a history of significant depression or drug abuse
* Volitional movements present during EMG testing in bilateral lower extremities
* Unhealed spinal fracture
* Presence of significant contracture with loss of greater than two-thirds range of motion
* Presence of pressure ulcers
* Current Pregnancy

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2029-04-15 (Estimated); Study Completion 2029-04-15 (Estimated)

PRIMARY OUTCOMES:
Safety of epidural spinal cord stimulator in chronic cervical patients | 1 year
  Incidence of adverse events (AEs) and serious adverse events (SAEs) including hypotension, other hemodynamic instability, infection, bleeding, significant pain, spasticity, or cerebrospinal fluid leak.

SECONDARY OUTCOMES:
Changes in blood pressure | 1 year
  Measured on tilt table testing. Both systolic and diastolic pressure will be assessed
Changes in heart rate | 1 year
  Measured on tilt table testing
Cognitive function | 1 year
  Measured using N-back testing
Cerebral blood flow | 1 year
  Measured using transcranial doppler
Muscle Sympathetic Nerve Activities (MSNA) | 1 year
  Microneurolography

OTHER OUTCOMES:
Volitional function on electromyography (EMG) | 1 year
  Using the modified brain motor control assessment (mBMCA) and electromyography (EMG).
Hand function | 1 year
  The Graded Redefined Assessments of Strength, Sensibility, and Prehension (GRASSP) functional score
Truncal stability | 1 year
  Using the modified Functional reach test (mFRT)
Stimulation settings optimization | 1 year
  Using Bayesian process

CONTACTS AND LOCATIONS:
Overall Officials: Ann Parr, MD, PhD, Principal Investigator — University of Minnesota; Manda Keller-Ross, PhD, DPT, PT, Principal Investigator — University of Minnesota; Nadine Mansour, MD, MPH, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be deposited in the Data Repository for the University of Minnesota (DRUM), an open-access institutional repository. Data stored during the project will be maintained in Box Secure Storage and REDCap before long-term archiving in DRUM.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Data will be shared after publication of the primary results and will remain available for at least 10 years, in accordance with the University of Minnesota's DRUM repository policies.
Access Criteria: Data will be openly accessible through DRUM without restrictions.
URL: https://hdl.handle.net/11299/166578